CLINICAL TRIAL: NCT05198999
Title: Aquatic-based Plyometric Exercises for Children With Hemiparetic Cerebral Palsy: A Randomized Controlled Study Investigating Effects on Postural Control and Functional Performance
Brief Title: Aquatic-based Explosive Strength Training in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0018/0069
Record Dates: First submitted 2021-12-19; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy
Keywords: Unilateral Cerebral Palsy; Balance; Rehabilitation; Exercise; Function; Activity; Participation
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Intervention Model Description: A prospective pre-test post-test randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aqua-PLYO group (Experimental): Participants in this group received the Aqua-PLYO training program
  Interventions: Other: Aquatic-based Plyometric Exercises
- Control group (Active Comparator): Participants in this group received the standard physical rehabilitation program
  Interventions: Other: Standard Physical Therapy

INTERVENTIONS:
Other: Aquatic-based Plyometric Exercises — The Aqua-PLYO group received the aquatic plyometric exercise training for 45 minutes, three times per week for 12 successive weeks. The training was conducted under close supervision of a licensed pediatric physical therapist according to safety performance guidelines defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association
  Arms: Aqua-PLYO group
Other: Standard Physical Therapy — The control group received the standard physical rehabilitation program conducted for 45 minutes, thrice a week for 12 consecutive weeks, and consisted of advanced balance training, gait training, postural and flexibility exercises, and strength training exercises.
  Arms: Control group

SUMMARY:
This study was designed to assess the effect of a 12-week aquatic-based plyometric (Aqua-PLYO) training on postural control and functional performance in children with hemiparetic cerebral palsy (h-CP). Fifty-six children with h-CP were randomly allocated to the Aqua-PLYO group (n = 28, received an Aqua-PLYO training program, trice/week, over 12 weeks) or the control group (n =28, received standard rehabilitation). Both groups were assessed for postural control and functional performance pre and post-treatment.

DETAILED DESCRIPTION:
Fifty-six children with h-CP were recruited from the Physical Therapy Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, King Khalid Hospital, and a tertiary referral hospital, Al-Kharj, Saudi Arabia. Their age ranged between 12 and 16 years, were functioning at levels I or II on the Gross Motor Function Classification System, and had spasticity level 1 or 1+ per the Modified Ashworth Scale. Children were excluded if they had fixed deformities, had leg-length discrepancy, underwent neuromuscular or orthopedic surgery in the last 12 months, submitted to BOTOX injection in the past 6 months, attentional neglect, cardiopulmonary problems preventing them from performing high-intense exercise training.

Outcome measures

1. Postural control: The dynamic limits of stability (LOSdynamic) indices were measured through the Balance Master system.
2. Functional performance: Functional performance was quantified using the 30-second sit-to-stand test (30sec-STS), Timed Up and Down Stairs test (TUDS), and the Dynamic Gait Index (DGI).

The Aqua-PLYO group received a 12-week Aqua-PLYO training, 45 minutes per session, three times a week for 12 consecutive weeks, in conformity with the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The Aqua-PLYO program consisted of ten unilateral and bilateral lower limb plyometrics in the form of hopping/bounding/jumping activities conducted in a water medium. The Aqua-PLYO training included a warm-up for 10 minutes and a cool-down for10 minutes. The control group received the usual physical therapy care, 45 minutes per session, three times a week for 12 consecutive weeks. The program consisted of advanced balance training, and gait training exercises, postural and flexibility exercises, strength training exercises.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparetic cerebral palsy
* Age between 12 to 16 years
* Spasticity level 1 or 1+ according to the Modified Ashworth Scale
* Gross motor function level I or II according to the Gross Motor Function Classification System

Exclusion Criteria:

* Structural deformities
* Musculoskeletal or neural surgery in the last year
* BOTOX injection in the last 6 months.
* Cardiopulmonary disorders limit the ability to engage in explosive exercise training
* Hemi-spatial neglect

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Directional Control | 2 months
  The amount of movement demonstrated in the desired direction, i.e. towards the target, to the amount of external movement in the opposite direction of the target, expressed as a percentage.
Reaction time | 2 months
  The time, taken by an individual to start shifting his center of gravity from the static position after the cue, measured in seconds
Movement Velocity | 2 months
  The average speed at which the center of gravity shifts, measured in degree/second
EndPoint Excursion | 2 months
  The distance willingly covered by the subject in his very first attempt towards the target, expressed as a percentage (%)
Maximum Excursion | 2 months
  The distance, the subject actually covered or moved his center of gravity toward a target, expressed as a percentage (%) of the dynamic limit of stability
Functional lower limb strength | 2 months
  the functional strength of lower limbs was measured by the 30-second sit-to-stand test. The test determines the number of sit-to-stand task repetitions performed within 30 seconds. The higher number of repetitions indicates better performance.
Functional mobility | 2 months
  Functional mobility was assessed by Timed Up and Down Stairs test. the test measures the time (second) that the subject takes to go upstairs, turn around, and come back down. Shorter time indicates better performance.
Gait balance | 2 months
  Gait balance was measured by the Dynamic Gait Index. The dynamic gait index quantified the ability of the participant to maintain walking balance while responding to different task demands, through various dynamic conditions.
  The index includes eight items, walking on level surfaces, changing speeds, head turns in horizontal and vertical directions, walking and turning 180 degrees to stop, stepping over and around obstacles, and stair ascent and descent.
  Each item is scored on a scale of 0 to 3, with 3 indicating normal performance and 0 representing severe impairment. The best possible score is 24. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University; Ragab K Elnaggar, PhD, Principal Investigator — Cairo University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No